CLINICAL TRIAL: NCT06630962
Title: Evaluating the Impact of Financial Navigation on Financial Catastrophe and Distress for Cancer Care: A Randomized Control Trial- COST-FIN
Brief Title: Evaluating the Impact of Financial Navigation on Financial Catastrophe and Distress for Cancer Care
Acronym: COST-FIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STU00221204
Record Dates: First submitted 2024-09-18; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Breast Neoplasm; Prostate Neoplasm; Colon Neoplasm; Rectal Neoplasm
Keywords: Financial Navigation; Financing Cancer Care; Nigeria; Breast Neoplasm; Prostate Neoplasm; Colon Neoplasm; Rectal Neoplasm; Health Insurance; Randomized Control Trial; Healthcare Cost; Health Expenditure; Financial Risk Sharing; Universal Health Insurance; National Health Insurance Scheme; Catastrophic Health Spending; Financial Distress; Sub-Saharan Africa; Health Plan Implementation; Global Health; Healthcare Economics and Organizations; Clinical Oncology; Cancer Care Facilities; Surgical Oncology; Global Burden of Disease; Social Determinants of Health; Health Impact Assessment
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Potential Crossover: An interim analysis will be conducted once 50% of the recruitment target (100 participants total) have completed at least 6-months of follow-up, which is estimated to occur at approximately 1 year from start of the study. If significant differences between the Financial Navigation Program (FNP) and routine care arms are observed, all enrolled participants in the control arm will be given access to the FNP. Endpoint-related data will be collected until study completion (1-year follow-up for all enrolled participants).
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Financial Navigation Arm (Experimental): A financial navigator will educate these participants on financial literacy, insurance plans and payment options available through charities and financial assistance programs. In addition to providing financial counseling, the financial navigator will verify participant insurance documents, maintain records of financial agreements, and coordinate payments with insurance companies.
  Interventions: Other: Financial Navigation Program
- Routine Care Arm (No Intervention): Participants will not have access to the services of the financial navigator. Financial counseling and assistance will be limited to what is routinely provided by the cancer center.

INTERVENTIONS:
Other: Financial Navigation Program — A salaried financial navigator will be hired by the study sites. All responsibilities of the navigator will revolve around the structured financial navigation program. There is currently no research indicating that such a role has been incorporated at cancer centers in sub-Saharan Africa.
  Through this program, the financial navigator will educate participants on financial literacy, insurance plans and payment options available through charities and financial assistance programs. In addition to providing financial counseling, the financial navigator will verify participant insurance documents, maintain records of financial agreements, and coordinate payments with insurance companies.
  Arms: Financial Navigation Arm

SUMMARY:
The goal of this study is to investigate the effectiveness of a structured financial navigation program in reducing financial catastrophe and financial distress for cancer patients in Nigeria.

The main study questions being investigated are:

1. If a financial navigation program can effectively and significantly reduce financial catastrophe and distress for cancer patients in Nigeria?
2. If a financial navigation program is financially sustainable and cost-effective for cancer centers in Nigeria?

Participants will be required to:

1. Complete surveys about their demographics, clinical history, and socioeconomic status
2. Complete questionnaires about their quality of life and psychological wellbeing
3. Report all costs related to their cancer care

Investigators will compare participants in the financial navigation program and those not in the financial navigation program to identify potential differences in catastrophic health expenditure and financial distress.

DETAILED DESCRIPTION:
Over 100,000 individuals are diagnosed with cancer annually in Nigeria, the highest burden out of all countries in sub-Saharan Africa (SSA). Treatment options are limited and often delayed due to lack of insurance coverage and high out-of-pocket costs, which is devastating for Nigeria's 83 million living in poverty (40% of the population). Importantly, it is estimated that 77-94% of cancer patients in SSA face financial catastrophe (FC) where health expenses exceed 25% of household expenditure, 40% of non-subsistence expenditures, or 10% of household income.

While Nigeria has recently planned to invest 300 billion USD in the National Cancer Control Plan, a comprehensive initiative to centralize and strengthen multidisciplinary cancer care, high-quality research on innovative methods to eliminate cost barriers and make treatment affordable is needed.

In the United States, structured financial navigation programs (FNP) have been successful in helping patients finance their cancer care, and save costs, and have been associated with reduced levels of financial distress. However, there is paucity of data high-quality on the effectiveness of an FNP for cancer care in SSA.

The proposed study will investigate the effectiveness of an FNP in reducing financial catastrophe and distress for cancer patients in Nigeria. The FNP will hire financial navigators (FNs) at the cancer centers to educate patients on financial literacy, enroll patients in insurance, and find alternative funding sources, such as charitable solutions. The randomized control trial will enroll 200 newly diagnosed breast, colorectal, or prostate cancer patients at two cancer centers in Lagos, Nigeria, and investigate the impact of the FNP on:

1. The incidence of financial catastrophe
2. Financial distress
3. Budget and financial sustainability analysis of the FNP -- by conducting a cost-effectiveness analysis by comparing the program's cost to the benefits in terms of funding secured and number of participants enrolled in insurance.

This study -- the first of its kind in SSA -- will inform the potential for FNPs to reduce the financial burden of cancer treatment in resource-constrained settings. If effective, programs like this would serve as an invaluable resource to increase access to care and in turn improve cancer outcomes in the region.

In light of Nigerian government's recently renewed interest in improving access to cancer care, findings from this study will be crucial in health policy reform. Further, this study's findings will inform and influence cancer care in SSA, and will prompt effectiveness in other similar contexts.

Finally, if found to be effective, data from this investigation will lay the foundation to support an R01-level study to comprehensively evaluate the implementation and adoption of FNPs in Nigeria and other parts of SSA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Recently diagnosed with breast, colorectal or prostate cancer within 6 weeks of presentation at the study site
* Have not received definitive chemotherapy, radiotherapy, or undergone major surgery (diagnostic or temporary interventions, such as excisional biopsy or temporary colostomy may still enroll)
* Candidate for definitive cancer treatment

Exclusion Criteria:

* Unable to provide consent
* Has initiated definitive cancer treatment at the study site or elsewhere in the past
* Only receiving best supportive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of financial catastrophe (FC) | From enrollment to 12 months
  To compare the incidence of FC between participants in the financial navigation program (FNP) and control arms.
  FC is defined as treatment-related costs that exceed 10% of household income (HHI), 25% of total household expenditure (HHE), or 40% of non-essential household spending (HSE). All direct and indirect out-of-pocket (OOP) costs of cancer care will be summed for each participant and represented as a proportion of HHI, HHE, and HSE.
Levels of financial distress (FD) | From enrollment to 3, 6 and 12 months
  To compare the levels of FD experienced between participants in the FNP and control arms.
  Financial Distress (FD) will be measured using the FACIT-COST tool, a validated patient-reported measure with scores ranging from 0-44 (higher scores represent better financial well-being). FACIT-COST scores will be assessed for all participants at 3, 6, and 12 months from enrollment, and mean scores at 6 months will be compared between both study arms.

SECONDARY OUTCOMES:
Rate of cost-related non-adherence | From enrollment to 6 months
  Exploratory analysis to compare the rates of treatment non-adherence related to treatment costs between the FNP and control arms.
  Data on adherence and reasons for non-adherence will be collected through structured interviews with participants and their treating medical oncologists 6 months post-enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Lumati, Principal Investigator — Northwestern University
Locations (2):
- Nigeria (2):
  - Obafemi Awolowo University Teaching Hospitals Complex, Ile-Ife
  - Lakeshore Cancer Center, Lagos

IPD SHARING:
Plan to Share IPD: Yes
Demographic, socioeconomic, clinical, cost, and patient-reported outcome data will be uploaded and shared for each enrolled participant. All data will be de-identified and dates will be excluded from the dataset.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be shared at study conclusion, once all analyses are complete. The data will be available to the wider research community indefinitely.
Access Criteria: Data will be accessible to anyone in the wider research community via the clinicaltrials.gov repository. The data will be identifiable through a unique identification code assigned by clinicaltrials.gov.

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] The Lancet. GLOBOCAN 2018: counting the toll of cancer. Lancet. 2018 Sep 22;392(10152):985. doi: 10.1016/S0140-6736(18)32252-9. Epub 2018 Sep 20. No abstract available. PMID 30264708
- [Background] Awodutire PO, Kolawole OA, Ilori OR. Data on the survival times of breast cancer patients in a Teaching Hospital, Osogbo. Data Brief. 2020 Aug 1;32:106109. doi: 10.1016/j.dib.2020.106109. eCollection 2020 Oct. PMID 32817870
- [Background] Ali-Gombe M, Mustapha MI, Folasire A, Ntekim A, Campbell OB. Pattern of survival of breast cancer patients in a tertiary hospital in South West Nigeria. Ecancermedicalscience. 2021 Feb 25;15:1192. doi: 10.3332/ecancer.2021.1192. eCollection 2021. PMID 33889201
- [Background] Gullickson C, Goodman M, Joko-Fru YW, Gnangnon FHR, N'Da G, Woldegeorgis MA, Buziba NG, Karugu C, Manraj SS, Lorenzoni CF, Hansen R, Finesse A, Somdyala NIM, Bukirwa P, Chingonzoh T, Chokunonga E, Liu B, Kantelhardt E, Parkin DM, Jemal A. Colorectal cancer survival in sub-Saharan Africa by age, stage at diagnosis and Human Development Index: A population-based registry study. Int J Cancer. 2021 Oct 15;149(8):1553-1563. doi: 10.1002/ijc.33715. Epub 2021 Jul 21. PMID 34164808
- [Background] Saluja S, Alatise OI, Adewale A, Misholy J, Chou J, Gonen M, Weiser M, Kingham TP. A comparison of colorectal cancer in Nigerian and North American patients: is the cancer biology different? Surgery. 2014 Aug;156(2):305-10. doi: 10.1016/j.surg.2014.03.036. Epub 2014 Jun 19. PMID 24953266
- [Background] Seraphin TP, Joko-Fru WY, Manraj SS, Chokunonga E, Somdyala NIM, Korir A, N'Da G, Finesse A, Wabinga H, Assefa M, Gnangnon F, Hansen R, Buziba NG, Liu B, Kantelhardt EJ, Parkin DM. Prostate cancer survival in sub-Saharan Africa by age, stage at diagnosis, and human development index: a population-based registry study. Cancer Causes Control. 2021 Sep;32(9):1001-1019. doi: 10.1007/s10552-021-01453-x. Epub 2021 Jul 10. PMID 34244896
- [Background] Ekeke O, Amusan O, Eke N. Management of prostate cancer in port harcourt, Nigeria: changing patterns. J West Afr Coll Surg. 2012 Jul;2(3):58-77. PMID 25452994
- [Background] Araghi M, Arnold M, Rutherford MJ, Guren MG, Cabasag CJ, Bardot A, Ferlay J, Tervonen H, Shack L, Woods RR, Saint-Jacques N, De P, McClure C, Engholm G, Gavin AT, Morgan E, Walsh PM, Jackson C, Porter G, Moller B, Bucher O, Eden M, O'Connell DL, Bray F, Soerjomataram I. Colon and rectal cancer survival in seven high-income countries 2010-2014: variation by age and stage at diagnosis (the ICBP SURVMARK-2 project). Gut. 2021 Jan;70(1):114-126. doi: 10.1136/gutjnl-2020-320625. Epub 2020 Jun 1. PMID 32482683
- [Background] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Background] Mustapha MI, Ali-Gombe M, Abdullahi A, Adenipekun A, Campbell OB. Financial Burden of Cancer on Patients Treated at a Tertiary Health Facility in South West Nigeria. J West Afr Coll Surg. 2020 Oct-Dec;10(4):23-29. doi: 10.4103/jwas.jwas_4_22. Epub 2022 Jun 8. PMID 35814963
- [Background] Sharma A, Alatise OI, Adisa AO, Arowolo OA, Olasehinde O, Famurewa OC, Omisore AD, Komolafe AO, Olaofe O, Katung AI, Ibikunle AD, Egberongbe AA, Olatoke SA, Agodirin SO, Adesiyun AO, Adeyeye A, Ibrahim K, Kolawole OA, Idris OL, Adejumobi MO, Ajayi AI, Olakanmi AO, Constable JC, Seier K, Gonen M, Brennan MF, Kingham TP. Treatment of colorectal cancer in Sub-Saharan Africa: Results from a prospective Nigerian hospital registry. J Surg Oncol. 2020 Feb;121(2):342-349. doi: 10.1002/jso.25768. Epub 2019 Nov 19. PMID 31742699
- [Background] Sharma A, Alatise OI, O'Connell K, Ogunleye SG, Aderounmu AA, Samson ML, Wuraola F, Olasehinde O, Kingham TP, Du M. Healthcare utilisation, cancer screening and potential barriers to accessing cancer care in rural South West Nigeria: a cross-sectional study. BMJ Open. 2021 Jul 26;11(7):e040352. doi: 10.1136/bmjopen-2020-040352. PMID 34312189
- [Background] Fapohunda A, Fakolade A, Omiye J, Afolaranmi O, Arowojolu O, Oyebamiji T, Nwogu C, Olawaiye A, Mutiu J. Cancer presentation patterns in Lagos, Nigeria: Experience from a private cancer center. J Public Health Afr. 2020 Dec 31;11(2):1138. doi: 10.4081/jphia.2020.1138. eCollection 2020 Dec 31. PMID 33623651
- [Background] Knapp GC, Wuraola FO, Olasehinde O, Romanoff A, Kingham PT, Alatise OI. The out-of-pocket cost of breast cancer care at a public tertiary care hospital in Nigeria: an exploratory analysis. Pan Afr Med J. 2022 Apr 5;41:272. doi: 10.11604/pamj.2022.41.272.24610. eCollection 2022. PMID 35784593
- [Background] Okoroh J, Sarpong DO, Essoun S, Riviello R, Harris H, Weissman JS. Does insurance protect individuals from catastrophic payments for surgical care? An analysis of Ghana's National Health Insurance Scheme at Korle-Bu teaching Hospital. BMC Health Serv Res. 2020 Jan 17;20(1):45. doi: 10.1186/s12913-020-4887-2. PMID 31952520
- [Background] Kasahun GG, Gebretekle GB, Hailemichael Y, Woldemariam AA, Fenta TG. Catastrophic healthcare expenditure and coping strategies among patients attending cancer treatment services in Addis Ababa, Ethiopia. BMC Public Health. 2020 Jun 22;20(1):984. doi: 10.1186/s12889-020-09137-y. PMID 32571275
- [Background] Alawode GO, Adewole DA. Assessment of the design and implementation challenges of the National Health Insurance Scheme in Nigeria: a qualitative study among sub-national level actors, healthcare and insurance providers. BMC Public Health. 2021 Jan 11;21(1):124. doi: 10.1186/s12889-020-10133-5. PMID 33430837
- [Background] GBD 2019 Universal Health Coverage Collaborators. Measuring universal health coverage based on an index of effective coverage of health services in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1250-1284. doi: 10.1016/S0140-6736(20)30750-9. Epub 2020 Aug 27. PMID 32861314
- [Background] Adisa AO, Lawal OO, Adesunkanmi AR. Paradox of wellness and nonadherence among Nigerian women on breast cancer chemotherapy. J Cancer Res Ther. 2008 Jul-Sep;4(3):107-10. doi: 10.4103/0973-1482.42640. PMID 18923201
- [Background] Okoronkwo IL, Ejike-Okoye P, Chinweuba AU, Nwaneri AC. Financial barriers to utilization of screening and treatment services for breast cancer: an equity analysis in Nigeria. Niger J Clin Pract. 2015 Mar-Apr;18(2):287-91. doi: 10.4103/1119-3077.151070. PMID 25666009
- [Background] ACTION Study Group; Kimman M, Jan S, Yip CH, Thabrany H, Peters SA, Bhoo-Pathy N, Woodward M. Catastrophic health expenditure and 12-month mortality associated with cancer in Southeast Asia: results from a longitudinal study in eight countries. BMC Med. 2015 Aug 18;13:190. doi: 10.1186/s12916-015-0433-1. PMID 26282128
- [Background] Sullivan R, Alatise OI, Anderson BO, Audisio R, Autier P, Aggarwal A, Balch C, Brennan MF, Dare A, D'Cruz A, Eggermont AM, Fleming K, Gueye SM, Hagander L, Herrera CA, Holmer H, Ilbawi AM, Jarnheimer A, Ji JF, Kingham TP, Liberman J, Leather AJ, Meara JG, Mukhopadhyay S, Murthy SS, Omar S, Parham GP, Pramesh CS, Riviello R, Rodin D, Santini L, Shrikhande SV, Shrime M, Thomas R, Tsunoda AT, van de Velde C, Veronesi U, Vijaykumar DK, Watters D, Wang S, Wu YL, Zeiton M, Purushotham A. Global cancer surgery: delivering safe, affordable, and timely cancer surgery. Lancet Oncol. 2015 Sep;16(11):1193-224. doi: 10.1016/S1470-2045(15)00223-5. PMID 26427363
- [Background] McKenzie F, Zietsman A, Galukande M, Anele A, Adisa C, Cubasch H, Parham G, Anderson BO, Abedi-Ardekani B, Schuz J, Dos Santos Silva I, McCormack V. African Breast Cancer-Disparities in Outcomes (ABC-DO): protocol of a multicountry mobile health prospective study of breast cancer survival in sub-Saharan Africa. BMJ Open. 2016 Aug 23;6(8):e011390. doi: 10.1136/bmjopen-2016-011390. PMID 27554102
- [Background] Bell-Brown A, Watabayashi K, Delaney D, Carlos RC, Langer SL, Unger JM, Vaidya RR, Darke AK, Hershman DL, Ramsey SD, Shankaran V. Assessment of financial screening and navigation capabilities at National Cancer Institute community oncology clinics. JNCI Cancer Spectr. 2023 Aug 31;7(5):pkad055. doi: 10.1093/jncics/pkad055. PMID 37561111
- [Background] Yezefski T, Steelquist J, Watabayashi K, Sherman D, Shankaran V. Impact of trained oncology financial navigators on patient out-of-pocket spending. Am J Manag Care. 2018 Mar;24(5 Suppl):S74-S79. PMID 29620814
- [Background] Edward JS, McLouth LE, Rayens MK, Eisele LP, Davis TS, Hildebrandt G. Coverage and Cost-of-Care Links: Addressing Financial Toxicity Among Patients With Hematologic Cancer and Their Caregivers. JCO Oncol Pract. 2023 May;19(5):e696-e705. doi: 10.1200/OP.22.00665. Epub 2023 Mar 8. PMID 36888937
- [Background] Doherty MJ, Thom B, Gany F. Evidence of the Feasibility and Preliminary Efficacy of Oncology Financial Navigation: A Scoping Review. Cancer Epidemiol Biomarkers Prev. 2021 Oct;30(10):1778-1784. doi: 10.1158/1055-9965.EPI-20-1853. Epub 2021 Aug 2. PMID 34341051
- [Background] Sadigh G, Gallagher K, Obenchain J, Benson A 3rd, Mitchell E, Sengupta S, Carlos RC. Pilot Feasibility Study of an Oncology Financial Navigation Program in Brain Cancer Patients. J Am Coll Radiol. 2019 Oct;16(10):1420-1424. doi: 10.1016/j.jacr.2019.07.014. No abstract available. PMID 31585660
- [Background] Shankaran V, Leahy T, Steelquist J, Watabayashi K, Linden H, Ramsey S, Schwartz N, Kreizenbeck K, Nelson J, Balch A, Singleton E, Gallagher K, Overstreet K. Pilot Feasibility Study of an Oncology Financial Navigation Program. J Oncol Pract. 2018 Feb;14(2):e122-e129. doi: 10.1200/JOP.2017.024927. Epub 2017 Dec 22. PMID 29272200
- [Background] Kircher SM, Yarber J, Rutsohn J, Guevara Y, Lyleroehr M, Alphs Jackson H, Walradt J, Desai B, Mulcahy M, Kalyan A, Benson AB, Agulnik M, Mohindra N, DeSouza J, Garcia SF. Piloting a Financial Counseling Intervention for Patients With Cancer Receiving Chemotherapy. J Oncol Pract. 2019 Mar;15(3):e202-e210. doi: 10.1200/JOP.18.00270. Epub 2019 Jan 9. PMID 30625023
- [Background] Watabayashi K, Steelquist J, Overstreet KA, Leahy A, Bradshaw E, Gallagher KD, Balch AJ, Lobb R, Lavell L, Linden H, Ramsey SD, Shankaran V. A Pilot Study of a Comprehensive Financial Navigation Program in Patients With Cancer and Caregivers. J Natl Compr Canc Netw. 2020 Oct 1;18(10):1366-1373. doi: 10.6004/jnccn.2020.7581. Print 2020 Oct. PMID 33022646
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Sadigh G, Coleman D, Lava N, Switchenko J, Vargas D, Duszak R Jr, Carlos RC. Patient-Specific Out-of-Pocket Cost Communication and Remote Financial Navigation in Patients with Multiple Sclerosis: A Randomized Controlled Feasibility Study. Mult Scler Relat Disord. 2022 Jun;62:103797. doi: 10.1016/j.msard.2022.103797. Epub 2022 Apr 10. PMID 35429820
- [Background] Sadigh G, Coleman D, Switchenko JM, Hopkins JO, Carlos RC. Treatment out-of-pocket cost communication and remote financial navigation in patients with cancer: a feasibility study. Support Care Cancer. 2022 Oct;30(10):8173-8182. doi: 10.1007/s00520-022-07270-5. Epub 2022 Jul 7. PMID 35796885
- [Background] Okoroh J, Essoun S, Seddoh A, Harris H, Weissman JS, Dsane-Selby L, Riviello R. Evaluating the impact of the national health insurance scheme of Ghana on out of pocket expenditures: a systematic review. BMC Health Serv Res. 2018 Jun 7;18(1):426. doi: 10.1186/s12913-018-3249-9. PMID 29879978
- [Background] Okoroh JS, Chia V, Oliver EA, Dharmawardene M, Riviello R. Strengthening Health Systems of Developing Countries: Inclusion of Surgery in Universal Health Coverage. World J Surg. 2015 Aug;39(8):1867-74. doi: 10.1007/s00268-015-3031-7. PMID 25802236
- [Background] Chakraborty NM, Fry K, Behl R, Longfield K. Simplified Asset Indices to Measure Wealth and Equity in Health Programs: A Reliability and Validity Analysis Using Survey Data From 16 Countries. Glob Health Sci Pract. 2016 Mar 25;4(1):141-54. doi: 10.9745/GHSP-D-15-00384. Print 2016 Mar. PMID 27016550
- [Background] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Background] Nwankwo T, Ogunyemi AO, Maduafokwa BA, Isikekpei BC, Alabi AO, Adegboyega BC, Otokpa E. Psychosocial Support and Cost Burden of Cancer Among Patients Attending Tertiary Oncology Clinics in Lagos State, Nigeria. Asian Pac J Cancer Prev. 2023 Jul 1;24(7):2313-2319. doi: 10.31557/APJCP.2023.24.7.2313. PMID 37505761
- [Background] Shih W. Problems in dealing with missing data and informative censoring in clinical trials. Curr Control Trials Cardiovasc Med. 2002 Jan 8;3(1):4. doi: 10.1186/1468-6708-3-4. PMID 11985778
- [Background] DeSouza CM, Legedza AT, Sankoh AJ. An overview of practical approaches for handling missing data in clinical trials. J Biopharm Stat. 2009 Nov;19(6):1055-73. doi: 10.1080/10543400903242795. PMID 20183464
- [Derived] Sohail AH, Afolaranmi O, Wuraola FO, Caputo M, Guiterrez G, Oyewole A, Ebekue DO, Adegbite ZO, Awe C, Ogunniyi T, Opeyemi A, Nwankwo C, Uwechue F, Sherman D, Lambert CN, Adedayo J, Diaz K, Christian EN, Abdulkareem F, Akin-Adigun O, Akingbola A, Okeke S, Knapp G, Dare A, Aduloju T, Akinwumi M, Kohli-Lynch CN, Chen R, Nwogu C, Hirschhorn LR, Adin-Cristian A, Iwuji C, Ilegbune O, Jimoh M, Chugani B, Oputa O, Murthy S, French D, Ackermann R, Murphy R, Seddoh A, Kingham P, Alatise OI, Lumati JS. Evaluating the Impact of Financial Navigation on Financial Catastrophe and Distress for Cancer Care: A Randomized Control Trial- COST-FIN. Res Sq [Preprint]. 2026 Jan 21:rs.3.rs-7686399. doi: 10.21203/rs.3.rs-7686399/v1. PMID 41646304
- [Derived] Sohail AH, Afolaranmi O, Wuraola FO, Caputo M, Gutierrez G, Oyewole A, Ebekue DO, Adegbite ZO, Awe C, Ogunniyi T, Opeyemi A, Nwankwo C, Uwechue F, Sherman D, Lambert CN, Adedayo J, Diaz K, Christian EN, Abdulkareem F, Akin-Adigun O, Akingbola A, Okeke S, Knapp G, Dare A, Aduloju T, Akinwumi M, Kohli-Lynch CN, Chen R, Nwogu C, Hirschhorn LR, Adin-Cristian A, Iwuji C, Ilegbune O, Jimoh M, Chugani B, Oputa O, Murthy S, French D, Ackermann R, Murphy R, Seddoh A, Kingham P, Alatise OI, Lumati JS. Evaluating the impact of financial navigation on financial catastrophe and distress for cancer care: a randomized control trial-COST-FIN. Trials. 2026 Jan 28. doi: 10.1186/s13063-026-09480-2. Online ahead of print. PMID 41606671
- See also: Partner site listing related materials to our study and patient enrollment — https://www.argo-research.org/cancer-clinical-trial/

DOCUMENTS (3):
  • Study Protocol (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT06630962/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-06): https://cdn.clinicaltrials.gov/large-docs/62/NCT06630962/SAP_001.pdf
  • Informed Consent Form (2024-04-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT06630962/ICF_002.pdf